CLINICAL TRIAL: NCT06025526
Title: Effectiveness of the Aktivplan Digital Intervention for Supporting Regular Heart-healthy Levels of Physical Activity Following Completion of a Phase II Rehabilitation Programme: a Clinical Pilot Study
Brief Title: Effectiveness of the Aktivplan Digital Intervention (ACTIVE-CaRe Pilot)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig Boltzmann Institute for Digital Health and Prevention (Other)
Collaborators: REHA Zentrum Salzburg (Unknown); Reha-Klinik Montafon (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23_5 ACTIVE-CaRe Pilot
Record Dates: First submitted 2023-08-23; First posted 2023-09-06 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Rehabilitation; Secondary Prevention; Cardiovascular Diseases
Keywords: Digital Health; Mobile Health; Electronic health; Smartphone App
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Other: aktivplan
- Control (Other)
  Interventions: Other: Usual care

INTERVENTIONS:
Other: aktivplan — The aktivplan digital intervention consists of a digital planning calendar for regular heart-healthy physical activity Towards the end of rehabilitation phase II, health professionals introduce aktivplan and plan a personalised physical activity plan together with their patients using shared decision-making. The physical activity plan is devised for the time after discharge from cardiac rehabilitation.
  In the aktivplan smatphone app, the patient can view their personalised physical activity plan, check off completed activities, enter additional unplanned activities, and open short videos with exercise instructions.
  Additional functions of aktivplan include patient-centered goal-setting, automated messages to the patient (motivational messages and reminders), and the possibility for health professionals to monitor all their patients' adherence to the physical activity plan and to contact individual patients directly via the app.
  Arms: Intervention
Other: Usual care — Usual care (standard of care) according to international and national cardiac rehabilitation guidelines.
  Arms: Control

SUMMARY:
The goal of this clinical pilot / feasibility study is to determine the feasibility of conducting a large-scale clinical effectiveness trial of the aktivplan digital intervention in cardiac rehabilitation patients.

The main questions this study aims to answer are:

* Is it feasible to conduct a large-scale (fully powered) effectiveness trial of the aktivplan digital intervention?
* What is the usability, user experience and user acceptance of the aktivplan digital intervention?

Patients enrolled in a phase II cardiac rehabilitation programme will be randomly allocated to either the intervention group (aktivplan digital intervention) ot the usual care control group and followed-up for 10 weeks after discharge from cardiac rehabilitation.

Patients in the intervention group will be given the aktivplan application (app) on their smartphone. A rehabilitation professional will plan a personalised heart-healthy physical activity plan together with the patient and enter it to the aktivplan app. The patient will be asked to follow their personal physical activity plan for 10 weeks, using the aktivplan app to document completed physical activity sessions.

Patients in the control group will receive the usual standard of care without the aktivplan digital intervention.

Researchers will analyse information such as the rate of recruitment, participant attrition, data completeness and technical stability of the app to determine the feasibility of conducting a large-scale clinical effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment to a cardiac rehabilitation programme phase II, or a rehabilitation programme phase II due to non-cardiac indication but displaying cardiovascular risk factors
* Ownership and use of a smartphone compatible with the aktivplan digital intervention and with internet connection
* Agreement to attend the study follow-up visit
* Written informed consent to take part in the study

Exclusion Criteria:

* Existing use of a digital intervention for regular heart-healthy physical activity
* Medical contraindications for incremental cycle ergometry test
* Medical contraindications for regular heart-healthy physical activity and sports
* Medical contraindications for use of a smartphone
* Inability to carry out cardiovascular training (e.g., due to significant musculoskeletal restrictions)
* Participation in another clinical study within the past 6 months
* Addiction or other medical conditions causing reduced decisional capacity
* Pregnant women in the third trimester
* Pregnant women in the first and second trimester with medical contraindication for physical activity and sports
* Breastfeeding women with medical contraindication for physical activity and sports
* Indication that patient is unlikely to follow study procedures (limited cooperation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 10 weeks
  Number of recruits per week
Drop-out rate | 10 weeks
  Number of drop-outs in at the 10-week follow-up visit
Data completeness | 10 weeks
  Percentage of missing data fields in the study database
Adherence to the aktivplan digital intervention | 10 weeks
  Automated usage logging of the aktivplan mobile application (Matomo platform)
Usability of the aktivplan digital intervention | 10 weeks
  mHealth App Usability Questionnaire (MAUQ)
User experience of the aktivplan digital intervention | 10 weeks
  AttrakDiff Short Questionnaire
User acceptance of the aktivplan digital intervention | 10 weeks
  Mobile Application Rating Scale (MARS)
Technical stability of the aktivplan digital intervention | 10 weeks
  Number and types of technical problems (qualitative data)
Use of alternative and additional strategies for supporting physical activity | 10 weeks
  Number and types of additional strategies (qualitative data)
Experiences and perspectives of patients regarding their study participation | 10 weeks
  Qualitative data from semi-structured interviews
Experiences and perspectives of rehabilitation professionals regarding the intervention and study procedures | 10 weeks
  Qualitative data from focus groups

SECONDARY OUTCOMES:
Exercise capacity | 10 weeks
  Incremental cycle ergometry test
Physical activity behaviour | 10 weeks
  Moderate to vigorous physical activity (MVPA)
Weight | 10 weeks
  Weight in kg
Blood pressure | 10 weeks
  Blood pressure in mmHg
Blood cholesterol | 10 weeks
  Total cholesterol, HDL-cholesterol, non-HDL-cholesterol, total cholesterol / HDL-cholesterol ratio
HbA1c | 10 weeks
  HbA1c level
Smoking | 10 weeks
  Number and type of smoking products per week (qualitative data)
Health-related quality of life | 10 weeks
  EQ-5D-5L Questionnaire
Exercise self-efficacy | 10 weeks
  Exercise Self-Efficacy Scale (ESES)
Patient safety | 10 weeks
  Adverse events reporting (number and severity of adverse events) assessed by the Medical Device Coordination Group (MDCG) form

CONTACTS AND LOCATIONS:
Overall Officials: Stefan T Kulnik, PhD MRes, Study Chair — Ludwig Boltzmann Institute for Digital Health and Prevention
Locations (2):
- Austria (2):
  - REHA Zentrum Salzburg, Salzburg, Salzburg
  - Reha-Klinik Montafon, Schruns, Vorarlberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leysen D, Reich B, Carrozzo AE, Crutzen R, Grote V, Kumar D, Mayr B, Niebauer J, Pfannerstill F, Propst EM, Wurhofer D, Sareban M, Smeddinck JD, Treff G, Kulnik ST. Feasibility of the aktivplan Digital Health Intervention for Regular Physical Activity Following Phase II Rehabilitation: Protocol for a Mixed Method Randomized Controlled Pilot Study (ACTIVE-CaRe Pilot). JMIR Res Protoc. 2025 Sep 15;14:e73704. doi: 10.2196/73704. PMID 40953438